CLINICAL TRIAL: NCT07211529
Title: Perioperative Paravertebral Block Reduces Postoperative Complications in Thoracic Surgery: An Observational Study
Brief Title: Intraoperative Paravertebral Block and Postoperative Complications
Acronym: IPVB and POCs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, GUO jiateng, Master of Clinical Medicine, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TJ-JRB202508092; TJ-JRB202508092 (Registry Identifier: Medical Ethics Committee of Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology)
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Video-assisted Thoracoscopic Surgery (VATS); Lung Cancer (Diagnosis); Pulmonary Infections; Respiratory Failure Without Hypercapnia; Pleural Effusion Due to Another Disorder (Disorder); Atelectasis; Bronchospasm; Pneumothorax; Pulmonary Embolism (Diagnosis); Bronchopleural Fistula; Acute Respiratory Distress Syndrome (ARDS)
Keywords: Paravertebral Block (PVB); Video-Assisted Thoracoscopic Surgery (VATS); Postoperative Complications
MeSH Terms: conditions — Lung Neoplasms; Disease; Respiratory Insufficiency; Pulmonary Atelectasis; Bronchial Spasm; Pneumothorax; Pulmonary Embolism; Respiratory Distress Syndrome; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: This study is designed as an observational investigation combining both retrospective and prospective components, focusing on patients undergoing thoracic surgery, primarily pulmonary and mediastinal procedures.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paravertebral Block (PVB)Group (Experimental): Participants in this arm will receive a paravertebral nerve block (PVB) performed intraoperatively under ultrasound guidance prior to the thoracic surgical procedure. The block will target the relevant thoracic vertebral levels corresponding to the surgical site. Standard local anesthetic agents will be administered according to institutional protocols. This intervention aims to provide perioperative analgesia, reduce postoperative pain, and potentially decrease the incidence of postoperative complications. All participants will also receive standard intraoperative monitoring and anesthesia management as per routine clinical practice.
  Interventions: Procedure: Paravertebral Block (PVB)
- Control Group (No Intervention): Participants in this arm will receive standard perioperative analgesia without the administration of a paravertebral block. Pain management will follow institutional protocols, which may include systemic opioids, non-steroidal anti-inflammatory drugs (NSAIDs), or other conventional analgesic methods. All participants will undergo the thoracic surgical procedure under standard intraoperative monitoring and anesthesia management as per routine clinical practice. This arm serves as the control group for evaluating the clinical effects of intraoperative paravertebral block on postoperative pain and complication rates.

INTERVENTIONS:
Procedure: Paravertebral Block (PVB) — Participants in this arm will receive a paravertebral nerve block (PVB) performed intraoperatively under ultrasound guidance prior to the thoracic surgical procedure. The block will target the relevant thoracic vertebral levels corresponding to the surgical site. Standard local anesthetic agents will be administered according to institutional protocols. This intervention aims to provide perioperative analgesia, reduce postoperative pain, and potentially decrease the incidence of postoperative complications. All participants will also receive standard intraoperative monitoring and anesthesia management as per routine clinical practice.
  Other Names: PVB; Paravertebral Analgesia; Paravertebral Injection; Ultrasound-Guided Paravertebral Block (UG-PVB / US-PVB); Thoracic Paravertebral Block (TPVB); Paravertebral Nerve Block
  Arms: Paravertebral Block (PVB)Group

SUMMARY:
This study aims to evaluate the clinical association between intraoperative paravertebral block and the reduction of postoperative complications following thoracic surgery.

DETAILED DESCRIPTION:
This study is designed as an observational investigation combining both retrospective and prospective components, focusing on patients undergoing thoracic surgery, primarily pulmonary and mediastinal procedures.

Retrospective analysis: We will collect data from patients across multiple campuses of Tongji Hospital who previously underwent thoracic surgery with intraoperative paravertebral block. These cases will be retrospectively analyzed to explore the association between paravertebral block and the reduction of postoperative complications.

Prospective evaluation: For patients enrolled prospectively, we will collect perioperative biochemical parameters, including MMP3, neutrophils, leukocytes, PCT, CRP, and other relevant regulatory factors. Postoperative outcomes will be assessed by recording cough and pain scores, as well as time to first flatus and defecation at 24 and 48 hours after surgery. In addition, patients will be followed for 30 days to document the incidence of postoperative complications.

Clinical correlation: The association between the measured biomarkers and patient outcomes will be systematically evaluated to determine their clinical relevance in predicting prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 years or older.
2. Scheduled to undergo thoracic surgery via Video-Assisted Thoracoscopic Surgery (VATS) or Robotic-Assisted Thoracoscopic Surgery (RATS), including wedge resection, segmentectomy, lobectomy, or mediastinal surgery.
3. Signed informed consent obtained prior to study participation. -

Exclusion Criteria:

1. Patients who refuse to provide informed consent.
2. Anesthesiologists who have not received training in ultrasound-guided paravertebral block (PVB-US).
3. History of ipsilateral thoracic surgery.
4. Conversion to open thoracotomy during the procedure.
5. Patients who did not complete the scheduled surgery due to disease progression or medical reasons.
6. Patients who are lost to follow-up or refuse postoperative follow-up. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complications | 1 to 3 months postoperatively
  Postoperative complications following thoracic surgery will be assessed as the primary outcome. These complications include pulmonary infection, respiratory failure, pleural effusion, atelectasis, bronchospasm, pneumothorax, aspiration-induced lung injury, pulmonary embolism, bronchopleural fistula, and acute respiratory distress syndrome (ARDS). The incidence of these complications will be systematically recorded and analyzed to evaluate the clinical impact of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang qin Zhang, Principal Investigator — Huazhong keji daxue tongji yixue yuan fushu tongji yiyuan
Locations (1):
- Tongji Medical College of HUST: Huazhong University of Science and Technology Tongji Medical College Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-07-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT07211529/Prot_000.pdf